CLINICAL TRIAL: NCT06807944
Title: Association Between Salivary Soluble RANKL, OPG Concentration and Mandibular Resorption to Clinically Predict Severe Residual Ridge Resorption Risk
Status: Completed | Type: Observational
Sponsor: Nguyen Thu Thuy (Other)
Responsible Party: Sponsor-Investigator, Nguyen Thu Thuy, Assoc. Prof., DDS., PhD, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: 488/HĐĐĐ-DHYD
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Edentulism in Lower Jaw

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrophic mandibular ridge
- Non-Atrophic mandibular ridge

SUMMARY:
Background. Affecting all individuals, residual ridge resorption (RRR) is a prevalent, progressive condition developing post tooth loss, often remaining silent until denture instability occurs. The molecular mechanisms and predictive bone biomarkers for severe RRR in edentulous individuals are poorly understood.

Object.This study aimed to investigate:

1. The association between salivary soluble Receptor activator of nuclear factor-κB ligand (RANKL), osteoprotegerin (OPG) concentration and the extent of mandibular resorption
2. Propose a way to clinically predict severe RRR risk. Methods.This cross-sectional study, conducted at the Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City, Vietnam (November 2021 to April 2024), enrolled 140 systemically healthy, edentulous adults (mean age 69.2 ± 8 years). Participants were stratified into atrophic (n=70) and non-atrophic (n=70) groups based on mandibular height. Demographic data (age, sex), edentulous duration, and denture history were recorded. Unstimulated whole saliva samples (5 mL) were collected, and salivary RANKL and OPG concentrations were quantified by ELISA.

DETAILED DESCRIPTION:
This cross-sectional study was approved by the Ethical Committee Board of the University of Medicine and Pharmacy in Ho Chi Minh City (UMP) (No.488/HĐĐĐ-ĐHYD), recruited participants between November 2021 and April 2024. All participants provided informed and written consent before clinical examinations and saliva. A convenience sampling method was employed. Of the 254 potential edentulous participants, 140 participants were included in the study.

Participant grouping: Participants underwent panoramic radiography to assess mandibular ridge height. They were classified into two groups. Atrophic groups have mandibular ridge heights less than 25 mm anteriorly and less than 16 mm posteriorly. In the non-atrophic group, mandibular ridge height is ≥ 25 mm anteriorly and ≥ 16 mm posteriorly.

Clinical factors: The participant's age, sex, duration of edentulism, and past complete denture experience were collected by the patient or patient's relative interview.

To obtain unstimulated whole saliva from each participants, approximately 5 ml was collected. Before the collection, all participants were instructed to refrain from eating and drinking for at least 30 minutes. Between 7:00 and 8:00 a.m., the collection was conducted through expectoration into sterile polypropylene tubes. Immediately after collection, the samples were placed in a cool box containing an ice pack and then hand-delivered to the Center for Molecular Biomedicine at UMP, Ho Chi Minh City, Vietnam.

RANKL and OPG salivary levels were measured using enzyme-linked immunosorbent assay Data analysis, including the relationship between RANKL, OPG and other variables, and the development of a predictive nomogram for high-risk bone resorption, was performed using R language version 3.4.0.

ELIGIBILITY:
Inclusion Criteria:

* complete edentulism for more than 3 years
* age > 35 years old
* no history of bone augmentation or mandibular defects

Exclusion Criteria:

* systemic diseases known to affect bone metabolism or immune function
* a history of malignancy
* salivary gland disease
* using antibiotics or immunosuppressant medications within 3 months

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Edentulous participants seeking oral care and treatment at the Faculty of Dentistry Clinic of the University of Medicine and Pharmacy Ho Chi Minh City from November 2021 to April 2024.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The concentration level of nuclear factor-κB ligand (RANKL) | within 6 months after sample collection
  It is measured using enzyme-linked immunosorbent assay (ELISA) kits (CSBE05125h, Cusabio, China ) mixing with the participant saliva
The concentration level of osteoprotegerin (OPG) | within 6 months after sample collection
  It is measured using enzyme-linked immunosorbent assay (ELISA) kits (CEHTNFRSF11B, Invitrogen, Massachusetts, USA ) mixing with the participant saliva

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Medicine and Pharmacy Ho Chi Minh City, Viet Nam, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Privacy concern